CLINICAL TRIAL: NCT05508633
Title: The Instant Efficacy and Safety of Alverine in Decreasing Portal Hypertension: an Exploratory Pilot Study
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, department of gastroenterology, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZXH2022002.01
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Portal Hypertension
Keywords: Portal hypertension; Alverine
MeSH Terms: conditions — Hypertension, Portal | interventions — alverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Alverine (Experimental): Alverine 60mg (1 capsule), orally
  Interventions: Drug: Alverine Citrate
- High dose Alverine (Experimental): Alverine 120mg (2 capsules), orally
  Interventions: Drug: Alverine Citrate

INTERVENTIONS:
Drug: Alverine Citrate — Low-dose group: Alverine (60 mg, 1 capsule) High-dose group: Alverine (120 mg, 2 capsules) The drug is orally given with 200 ml warm water after measurement of the baseline portal pressure.

SUMMARY:
The main purpose of this exploratory study was to investigate the instant efficacy and safety of alverine oral administration in decreasing portal hypertension.

Condition of disease: Cirrhotic portal hypertension

Intervention/treatment:

Drug: Alverine 60 mg (1 capsule), orally Drug: Alverine 120 mg (2 capsules), orally

DETAILED DESCRIPTION:
Portal hypertension is the main non-neoplastic consequence of chronic liver disease and represents the leading cause of death and liver transplantation in patients with liver cirrhosis. While no effective treatment has been addressed to cirrhosis, reduction of portal hypertension significantly prevents the complications of cirrhosis and then remarkedly improves patients' prognosis. At present, pharmacologic managements of portal hypertension recommended by guidelines are vasoactive modulators and nonselective β-blockers (NSBBs). Although these treatments are effective in reducing portal pressure in responsive patients, they are still far from ideal due to adverse events and unpredictable response. As the trends of death resulting from cirrhosis and portal hypertension remain high, the pathophysiology of portal hypertension needs to be further investigated, and novel therapeutic strategies for portal hypertension are needed urgently.

Alverine citrate is an antispasmodic drug with specific action on the smooth muscle of the alimentary tract and uterus, and does not affect the heart, blood vessels, or tracheal muscle at therapeutic doses. It was used in conditions such as irritable bowel syndrome, painful diverticular disease of the colon and primary dysmenorrhea to relief the smooth muscle spasm. Alverine citrate has been reported as a selective antagonist of serotonin receptor 1A (HTR1A) that reduced the visceral pronociceptive effect of serotonin. We found that alverine had the therapeutic potential on portal hypertension by selectively antagonizing HTR1A in preclinical animal models.

The trial aimed to evaluate the instant efficacy and safety of alverine oral administration in decreasing portal pressure of patients with cirrhotic portal hypertension.

The trial was planned as a single center prospective randomized investigation evaluating two doses of alverine on instant portal pressure reduction in 20 subjects two hours after receiving either high dose (120 mg) or low dose (60 mg) of alverine. The primary outcome measurement is the change in portal pressure from baseline to 2 hours after start of orally administration. Alverine response rate and safety will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Confirmed evidence of cirrhosis/ Cirrhosis diagnosed by liver biopsy or by imaging studies showing a nodular liver, splenomegaly and/or collateral.
3. Portal pressure greater than equal to (≥)10 mmHg.
4. Signed informed consent.

Exclusion Criteria:

1. Use of non-selective beta-blockers (e.g. carvedilol, propranolol) or statins within 1 month prior to dosing.
2. Moderate or massive ascites, overt hepatic encephalopathy, gastrointestinal bleeding and other complications within 1 week.
3. Previous splenectomy, cardia periesophageal vascular dissection, transjugular intrahepatic portosystemic shunt (TIPS), liver transplantation, etc.
4. Coagulopathy, including platelet count < 50× 10^9/ L, international normalized ratio (INR) of prothrombin time ≥1.5.
5. Serum total bilirubin ≥ 5 fold of upper limits of normal; serum sodium level < 125 mmol/ L; white blood cell count < 1× 10^9/ L.
6. Severe chronic renal insufficiency (eGFR (CKD-EPI) < 20 ml/min/1.73 m2).
7. Presence of hepatic vein, portal vein, splenic vein thrombosis or cavernous transformation of the portal vein.
8. Poorly controllable hypertension or diabetic patient; severe background disease like chronic respiratory failure, circulatory failure, kidney failure etc.
9. Clinically diagnosed or suspected as malignancy, including hepatocellular carcinoma.
10. Any uncontrolled active infection (e.g. lung infection, abdominal infection, HIV, etc) 4 weeks prior to enter in the study.
11. Patient who are allergy to the experimental drug.
12. Patients with abnormal mental symptoms or taking tricyclic antidepressants and similar drugs in the past 4 weeks.
13. Gestation or lactation period women and women who plan to get pregnant during the study period.
14. Patients who are participating other trials or have taken part in other in the past 4 weeks.
15. Other situation where PI thinks the patient should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in portal pressure | Change in portal pressure from baseline to 2 hours after start of orally administration
  Change in portal pressure from baseline to 2 hours after start of orally administration

SECONDARY OUTCOMES:
Treatment response rate | 2 hours
  The percentage of patients with portal pressure decreased by more than 10% fro baseline at 2h.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, Principal Investigator — Director of department of gastroenterology
Locations (1):
- Shanghai Changzheng hospital, Shanghai, Shanghai Municipality, China